CLINICAL TRIAL: NCT06178328
Title: 'Things You Do': An Observational Pilot Trial of a Brief Psychological Intervention Among People Seeking Online Mental Health Services
Brief Title: Observations of a Brief Online Psychological Intervention Among People Seeking Online Mental Health Services
Status: Recruiting | Type: Observational
Sponsor: University of Regina (Other)
Responsible Party: Sponsor
Other Study IDs: 414
Record Dates: First submitted 2023-11-30; First posted 2023-12-21 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Depression, Anxiety
Keywords: internet-delivered cognitive behaviour therapy; brief intervention
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Brief psychological intervention (Things You Do): All participants will have access to the online course materials for a period of 4 weeks from the time of enrolment. The materials are self-directed and can be accessed at any time during the 4-week period.
  Interventions: Behavioral: Things You Do Course

INTERVENTIONS:
Behavioral: Things You Do Course — Participants receiving the brief psychological intervention ('Things You Do' Course) will have access to a single online lesson that includes course materials and printable materials (i.e., an activity guide and planner) that can be retained for longer-term use. The course materials include an introduction to the purpose and content of the course, education about factors that impact mental health, and information about the 'Big Five' things participants can do to improve their mental health. Participants will also receive automated no-reply emails (5 days/week) through the intervention platform to remind them to practice the skills from the course.

SUMMARY:
Since 2012, the Online Therapy Unit has been offering Internet-delivered cognitive behaviour therapy (ICBT). ICBT represents a convenient method for individuals to access care for depression and anxiety. In ICBT, clients receive access to standardized lessons that provide the same information and skills as traditional face-to-face CBT. ICBT courses often span 6-12 weeks. There is now growing evidence that clients with symptoms of depression and anxiety can benefit from a single session brief intervention that offers practical strategies for improving mental health, but the investigators are uncertain about the interest in such a lesson among those seeking online mental health care. The Things You Do Course, therefore, is designed to provide clients with 5 key actions that clients can take to improve their emotional wellbeing.

In this study, the Online Therapy Unit (OTU) is examining how effective the Things You Do Course is in helping clients manage their symptoms of depression and anxiety and improve their emotional wellbeing. The OTU is also exploring the extent to which clients are satisfied with the course, and what factors contribute to improvements in symptoms, as measured by a number of questionnaires. The research will ultimately be used to improve how the OTU will deliver ICBT and to inform whether to include the single session course within existing online mental health service options.

DETAILED DESCRIPTION:
A scarcity of mental health care practitioners across Canada has resulted in extensive wait times. This issue is compounded by the significant cost associated with accessing psychological services, lack of awareness about service availability, and the constraints of time that hinder using long-term (multi-session) psychological therapies. These challenges are frequently cited as barriers to the access and utilization of psychological services in Canada. Unfortunately, this situation leaves many Canadians grappling with physical and mental disabilities, economic productivity losses, and facing an elevated risk of suicide due to unmet mental health care needs. Thus, there is a need for efficient and sustainable service delivery models that enable quick access to treatment for mental health concerns.

There is substantial evidence for the use of internet-delivered cognitive behaviour therapy (ICBT) as an alternative to face-to-face cognitive behaviour therapy (CBT) for the treatment of common mental health concerns such as anxiety and depression. The duration of ICBT courses varies, but most involve several lessons spanning 6-12 weeks. Offering brief, low-intensity supports may help alleviate barriers related to treatment seekers' time constraints.In face-to-face services, there is growing evidence that clients with symptoms of depression and anxiety can benefit from a single session intervention, but there is limited research on the use of single session interventions in ICBT, particularly within Canada.

Preliminary findings from the eCentre Clinic in Australia on a single lesson intervention (i.e., the 'Things You Do' course; TYD) are promising. The TYD is a single online lesson that provides psychoeducation about factors that contribute to mental health, as well as 5 target areas that clients can focus on to improve their mental health: realistic thinking, meaningful activities, goal setting, healthy routines, and social connections. Clients who completed the TYD reported significant improvements in depression and anxiety from pre- to post-treatment, with changes maintained at 12-week follow-up.

Given these promising preliminary findings, investigators propose to implement and evaluate the acceptability and short-term effects of a single-session intervention, the 'Things You Do' (TYD), in a Canadian context. The TYD is focused on everyday behaviours and actions that most people can choose to do, that is, it comprises modifiable behaviours which most people would recognize as important for mental health. It therefore has the potential to serve as a scalable, self-guided mental health intervention.

The following research questions will be evaluated:

1. What will be the uptake of the TYD course relative to other online mental health courses in the Online Therapy Unit?
2. What are the baseline demographic and clinical (e.g., severity levels of anxiety and depression symptoms) characteristics of individuals who sign up for the TYD?
3. How acceptable is the TYD in a Canadian context, as assessed via participants' ratings and feedback on likes and dislikes about the course content and process?
4. Will participating in TYD result in a clinically significant reduction in symptoms related to anxiety and depression and improvements in other measures administered?
5. What baseline demographic and clinical characteristics are related to outcomes post-treatment?
6. What percentage of TYD participants express interest in seeking out and enrolling in other online services offered by the Online Therapy Unit and how many individuals from other online services offered by the Online Therapy Unit subsequently enroll in TYD?

The study will begin with a pilot trial to examine research question 4. The intention is to collect more information if feasible to answer the other research questions related to uptake of the course, exploration of demographic and clinical characteristics of those who take the course, acceptability of the course and feedback on the course, relationship of demographic and clinical characteristics to outcomes and subsequent use of other services after taking the TYD course.

ELIGIBILITY:
Inclusion Criteria:

* Canadian resident;
* Aged 18 years or older;
* Seeking services for mental health concerns

Exclusion Criteria:

* Living outside of Canada
* Unable to read and understand English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This observational pilot trial explores aspects of the TYD course within an online routine care setting, a first-of-its-kind in Canada. Prospective participants will self-refer after learning about the course from advertisements, information on the Online Therapy Unit website, or from healthcare providers, community organizations, or others.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-11-17 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
The Things You Do Questionnaire - 21 item (TYD-Q) | Pre-treatment, 2 weeks (mid-treatment), 4 weeks (post-treatment), and 17 weeks (follow-up)
  A 21-item questionnaire that includes five scales (Realistic Thinking, Meaningful Activities, Goals and Plans, Healthy Habits, and Social Connections) to measure everyday behaviours that are linked to emotional wellbeing. Scores range from 0 to 84.
Patient Health Questionnaire (PHQ-9) | Pre-treatment, 2 weeks (mid-treatment), 4 weeks (post-treatment), and 17 weeks (follow-up)
  9-item measure of depression symptoms. Higher total scores indicate greater severity of depression. Scores range from 0 to 27.
Generalized Anxiety Disorder 7-Item (GAD-7) | Pre-treatment, 2 weeks (mid-treatment), 4 weeks (post-treatment), and 17 weeks (follow-up)
  7-item measure of anxiety symptoms. Higher total scores indicate greater severity of anxiety. Scores range from 0 to 21.

SECONDARY OUTCOMES:
Days out of role - 1 item | Pre-treatment, 4 weeks (post-treatment), and 17 weeks (follow-up)
  The functional impairment item from the longer Kessler Psychological Distress - 10 item Plus (K10+) scale to measure disability. Respondents are asked how many days they have been unable to work at all in the previous 4 weeks. Scores range from 0 to 28
Satisfaction with life scale (SWLS) | Pre-treatment, 4 weeks (post-treatment), and 17 weeks (follow-up)
  5-item measure of life satisfaction. Participants indicate how much they agree or disagree with each of the 5 items using a 7-point scale that ranges from 7 strongly agree to 1 strongly disagree. Scores range from 5 to 35
Feedback questions | 4 weeks (post-treatment)
  Closed-ended questions about treatment satisfaction; open-ended questions regarding suggestions of how to improve the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Heather Hadjistavropoulos, PhD, Principal Investigator — University of Regina
Locations (1):
- Online Therapy Unit- University of Regina, Regina, Saskatchewan, Canada

REFERENCES:
- [Background] Faber, S. C., Williams, M. T., Metzger, I. W., MacIntyre, M. M., Strauss, D., Duniya, C. G., ... & Goghari, V. M. (2023). Lions at the gate: How weaponization of policy prevents people of colour from becoming professional psychologists in Canada. Canadian Psychology.
- [Background] Hahmann, T.; Kumar, M.B. Unmet Health Care Needs during the Pandemic and Resulting Impacts among First Nations People Living Off Reserve, Métis and Inuit; Statistics Canada: Ottawa, ON, Canada, 2022; Available online: https://www150.statcan.gc.ca/n1/pub/45-28-0001/2022001/article/00008-eng.htm# (accessed on 3 January 2023).
- [Background] Khattar J, Griffith LE, Jones A, De Rubeis V, de Groh M, Jiang Y, Basta NE, Kirkland S, Wolfson C, Raina P, Anderson LN; Canadian Longitudinal Study on Aging (CLSA) Team. Symptoms of depression and anxiety, and unmet healthcare needs in adults during the COVID-19 pandemic: a cross-sectional study from the Canadian Longitudinal Study on Aging. BMC Public Health. 2022 Dec 1;22(1):2242. doi: 10.1186/s12889-022-14633-4. PMID 36456993
- [Background] Statistics Canada. Health Fact Sheets: Mental Health Care Needs, 2018; Catalogue No. 82-625-X; Statistics Canada: Ottawa, ON, Canada, 2019; Available online: https://www150.statcan.gc.ca/n1/en/pub/82-625-x/2019001/article/00011-eng.pdf (accessed on 10 August 2022)